CLINICAL TRIAL: NCT04996966
Title: Effect of Human Umbilical Cord-derived Mesenchymal Stem Cells on Non-cardiac Surgery-induced Lung Injury in Patients With Ischemic Heart Disease
Brief Title: Effect of Human Umbilical Cord-derived Mesenchymal Stem Cells on Non-cardiac Surgery-induced Lung Injury
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DFDA-001
Record Dates: First submitted 2021-07-14; First posted 2021-08-09 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Ischemic Heart Disease; Lung Injury; Non-cardiac Surgery
Keywords: human umbilical cord-derived mesenchymal stem cells; lung injury
MeSH Terms: conditions — Myocardial Ischemia; Lung Injury | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Placebo Comparator): In the control group, saline containing 2% albumin (2ml/kg) were intravenously injected to the patient immediately after the surgery and at day 3 after the surgery.
  Interventions: Other: saline
- MSCs injection (Experimental): In the MSCs injection group, 1×10^6/kg human umbilical cord-derived mesenchymal stem cells were intravenously injected to the patient immediately after the surgery and at day 3 after the surgery.
  Interventions: Biological: human umbilical cord-derived mesenchymal stem cells

INTERVENTIONS:
Biological: human umbilical cord-derived mesenchymal stem cells — In the MSCs injection group, 1×10^6/kg human umbilical cord-derived mesenchymal stem cells were intravenously injected to the patient immediately after the surgery and at day 3 after the surgery.
  Arms: MSCs injection
Other: saline — In the control group, saline containing 2% albumin (2ml/kg) were intravenously injected to the patient immediately after the surgery and at day 3 after the surgery.
  Arms: control

SUMMARY:
This study is an exploratory clinical study to observe the improvement of lung function before and after the treatment by human umbilical cord-derived mesenchymal stem cells, and the purpose is to evaluate the safety and effectiveness of human umbilical cord-derived mesenchymal stem cells on non-cardiac surgery-induced lung injury in patients with ischemic heart disease. The study is a randomized parallel controlled study. Patients receive a review of which main content includes symptom improvement, lung function improvement, and adverse events.

DETAILED DESCRIPTION:
This study is an exploratory clinical study to observe the improvement of lung function before and after the treatment by human umbilical cord-derived mesenchymal stem cells, and the purpose is to evaluate the safety and effectiveness of human umbilical cord-derived mesenchymal stem cells on non-cardiac surgery-induced lung injury in patients with ischemic heart disease.

The study is a randomized parallel controlled study. The research process is as follows: 1. Sixteen eligible patients with ischemic heart disease were recruited, fully informed, and signed a consent form, and randomly divided into placebo control group (n=8) or hUC-MSCs treatment group (n=8); 2. Knee replacement was performed under general anesthesia in both groups. In the cell therapy group, 1×10^6/kg human umbilical cord-derived mesenchymal stem cells were intravenously injected to the patient immediately after the surgery and at day 3 after the surgery. Before the operation, 6 hours, 3 days, 7days, 14 days, and 28 days after the MSCs injection, all patients receive a review of which main content includes symptom improvement, lung function improvement, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* The electrocardiogram showed T wave change and ST segment depression
* New York Heart Association (NYHA) Classification of cardiac function Ⅰ-Ⅱ level
* The patient who first time to receive knee replacement
* General anesthesia lasted about 2h
* Signed informed consent

Exclusion Criteria:

* Does not meet the above selection criteria
* Unable to sign the informed consent
* Patients with a malignant tumor, other serious systemic diseases, or psychosis
* Pregnancy, lactation, and those who are not pregnant but do not take effective contraceptives measures
* The patient with a history of an allergic reaction to biological products or drug
* The patient has any infectious diseases (including bacterial and viral infections)
* The patient with cardiac pacemaker implantation within 3 months prior to enrollment
* The patient who had a stroke within 6 months prior to enrollment
* Unable to comply with the agreed timetable of this study
* Patients who are participating in other clinical trials
* Others who are clinically considered unsuitable for this treatment.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
oxygenation index | Before the operation, 6 hours, 3days, and 7days after the MSCs injection
  The change in oxygenation index after the operation

SECONDARY OUTCOMES:
The value of arterial blood cLAC | Before the operation and 7days after the MSCs injection
  The change in arterial blood cLAC after the operation
The content of IL-1β | Before the operation and 7days after the MSCs injection
  The change in venous blood IL-1β after the operation
The content of IL-6 | Before the operation and 7days after the MSCs injection
  The change in venous blood IL-6 after the operation
The content of TGF-α | Before the operation and 7days after the MSCs injection
  The change in venous blood TGF-α after the operation
The content of HMGB1 | Before the operation and 7days after the MSCs injection
  The change in venous blood HMGB1 after the operation
The content of IL-10 | Before the operation and 7days after the MSCs injection
  The change in venous blood IL-10 after the operation
The content of B-type natriuretic peptide (BNP) | Before the operation and 7days after the MSCs injection
  The change in venous blood B-type natriuretic peptide after the operation
electrocardiogram | Before the operation, 7days, and 28 days after the MSCs injection
  The change in electrocardiogram after the operation
The average length of stay in hospital | The average length of stay in hospital
  The change in the length of stay in hospital between the two groups
The visual analog scale（VAS）score | Before the operation, 6 hours, 3 days, 7days, 14 days, and 28 days after the MSCs injection
  The change in VAS score after the operation，the minimum value is 0 and the maximum value is 10, the higher scores mean a worse outcome.
The hospital for special surgery (HSS) Knee Score | Before the operation, 7days, and 28 days after the MSCs injection
  The change in HSS Knee Score after the operation, the minimum value is 0 and the maximum value is 100, the higher scores mean a better outcome.
The New York Heart Association (NYHA) Functional Classification | Before the operation, 7days, 14 days, and 28 days after the MSCs injection
  The change in NYHA Functional Classification after the operation, the lowest level is Class I and the highest level is Class IV, the higher level mean a worse outcome.
The 36-Item Short Form Survey (SF-36) | Before the operation and 28 days after the MSCs injection
  The change in SF-36 after the operation, the minimum value is 40 and the maximum value is 850, the higher scores mean a better outcome.
The Hamilton Anxiety Scale | Before the operation, 7days, 14 days, and 28 days after the MSCs injection
  The change in degree of anxiety after the operation, the minimum value is 0 and the maximum value is 56, the higher scores mean a worse outcome.
The incidence of allergic reaction | Before the operation, 6 hours, 3 days, 7days, 14 days, and 28 days after the MSCs injection
  The allergic reaction after the MSCs injection
The body temperature | Before the operation, 6 hours, 3 days, 7days, 14 days, and 28 days after the MSCs injection
  The body temperature before and after the operation
The pulse rate | Before the operation, 6 hours, 3 days, 7days, 14 days, and 28 days after the MSCs injection
  The pulse rate before and after the operation
The respiration rate | Before the operation, 6 hours, 3 days, 7days, 14 days, and 28 days after the MSCs injection
  The respiration rate before and after the operation
The blood pressure | Before the operation, 6 hours, 3 days, 7days, 14 days, and 28 days after the MSCs injection
  The blood pressure before and after the operation
The content of C-reactive protein (CRP) | Before the operation and 7 days after the MSCs injection
  The change in venous blood CRP after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Xiangrui Wang, Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai Tongji University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No